CLINICAL TRIAL: NCT01420848
Title: The Effectiveness of the Auriculotherapy on Reducing Stress and Anxiety in Nursing Student: Randomized Clinical Trial
Brief Title: Auriculotherapy Effectiveness on Stress and Anxiety in Nursing Student
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonice Fumiko Sato Kurebayashi, Leonice Fumiko Sato Kurebayashi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SISNEP CAAE 0107.0.360.000-11
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-06

CONDITIONS: Stress; Anxiety
Keywords: stress disorders; anxiety disorders
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic | interventions — Auriculotherapy; Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auriculotherapy Group (Active Comparator): The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
  Two points were chosen to treat stress and anxiety (Shenmen and Brainstem).
  Interventions: Other: Auriculotherapy
- Placebo Group (Placebo Comparator): Auriculotherapy by sham, at the fist and outer ear points. These points aren't indicated for stress and anxiety.
  Interventions: Other: Placebo Group
- Control Group (No Intervention): Control Group didn't receive any treatment and was evaluated at the same time and the same way of interventions group

INTERVENTIONS:
Other: Auriculotherapy — Auriculotherapy stimulates points to achieve better emotional balance, mental and physiological.
  Other Names: Auricular acupuncture
  Arms: Auriculotherapy Group
Other: Placebo Group — They were evaluated at the baseline,twelve sessions and 15-day follow-up and received 12 sessions through the Fist and Outer ear points.
  Other Names: Sham Group
  Arms: Placebo Group

SUMMARY:
Single-blind randomized controlled trial aimed to assess stress and anxiety levels in Nursing School students of Beneficence Portuguese Hospital and review the effectiveness of true and placebo auriculotherapy.

DETAILED DESCRIPTION:
Although researches on stress have a strong focus on stress at work,it is very important the evaluation of the stress and its consequences in Nursing students. This allows to understand which stress factors experienced in a negative way could interfere on the adaptive success in school activities. Students can experience symptoms of the alarm phase of stress such as tachycardia, muscle tension, skin and cold extremities, and also the second phase of stress such as headache, sleepiness, irritability and difficulty concentrating. High levels of stress have a substantial effect on attention and can lead to errors, lack of concentration and fluctuations in the level of attention. The auriculotherapy may have an important role as a coping strategy for stress and anxiety. It is a fast, relatively simple, easily performed, safe and without major side effects.

ELIGIBILITY:
Inclusion Criteria:

* Average and high score by the List of Stress Symptoms
* Voluntary participation in the study
* Availability of time for submission to the sessions

Exclusion Criteria:

* Pregnancy
* Medical license or vacation during the period
* Low score of stress

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana M Prado, Principal Investigator — University of Sao Paulo; Leonice FS Kurebayashi, Study Director — University of Sao Paulo; Maria Julia P Silva, Study Chair — University of Sao Paulo
Locations (1):
- Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Giaponesi ANL, Leão ER. Auriculotherapy as an intervention to reduce stress reduction among the nursing team in intensive care. Nursing (São Paulo);12(139):575-579, dez. 2009. ilus.
- [Derived] do Prado JM, Kurebayashi LF, da Silva MJ. Efficacy of auriculotherapy for the reduction of stress in nursing students: a randomized clinical trial. Rev Lat Am Enfermagem. 2012 Jul-Aug;20(4):727-35. doi: 10.1590/s0104-11692012000400013. English, Portuguese, Spanish. PMID 22990158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of students was conducted between January and July 2011 at the Nursing School of Portuguese Beneficence Hospital. Eighty five people were invited and seventy one subjects were enrolled and randomized into 3 groups.
Pre-assignment Details: No sample size calculation was done for this study because the number of the population was small and it was decided to invite all students to attend nursing school test.
Groups:
- Auriculotherapy Group: The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
  Two points were chosen to treat stress and anxiety (Shenmen and Brainstem).
  Auriculotherapy : Auriculotherapy stimulates points to achieve better emotional balance, mental and physiological.
Period: Overall Study
Arm/Group | Auriculotherapy Group | Control Group | Placebo Group
Started | 24 | 25 | 22
Completed | 24 | 25 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy Group | Control Group | Placebo Group | Total
Number analyzed (Participants) | 24 | 25 | 22 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 22 | 71
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.21 (5.97) | 28.68 (6.57) | 30.91 (8.34) | 28.93 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 22 | 64
  Male | 4 | 3 | 0 | 7
Region of Enrollment [Number; unit: participants]
  Brazil | 24 | 25 | 22 | 71

OUTCOME MEASURES:

1. Primary Outcome: Students Stress Levels
Description: The List of Symptoms of Stress is an evaluation questionnaire which consists of a list of 59 psycho-physiological and psychosocial stress, in which the subject must associate to each symptom of the four answers: never (0), rarely (1 ), often (2) or always (3). The scores are added together and the answers provide the level of stress the individual.In this questionnaire to score from 0 to 11 is void, 12 to 29 (low level), 30 to 59 (medium level), 60 to 120 (high level) and 120 to 177, very high level. Participants below 29 points were excluded.
Time Frame: 90 days
Population: It was analysed only the subjects that ended the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy Group | Control Group | Placebo Group
Number analyzed (Participants) | 24 | 25 | 22
units on a scale | 75.62 (26.50) | 67.72 (22.38) | 72.45 (25.65)
Statistical Analysis 1: Comparison: Auriculotherapy Group vs Control Group vs Placebo Group; It was carried out the analysis of variance (ANOVA) among the groups at the 3rd (12 sessions) Hypothesis: there is at least one difference among the groups; Test type: Superiority or Other; p = 0.006, ANOVA — It was used the Post Hoc and the statistical significance was p<0.05
Statistical Analysis 2: Comparison: Auriculotherapy Group vs Control Group vs Placebo Group; It was verified the normality of data distribution and the homogeneity of variance. It was carried out the analysis of variance (ANOVA) among the groups at the follow-up (after 15 days); Test type: Superiority or Other; p = 0.023, ANOVA — The statistical significance was p<0.05

2. Secondary Outcome: Students Anxiety Levels
Description: The State-Trait Anxiety Inventory consists of 2 scales, each one containing 20 items. One of the scales evaluates state anxiety, characterized by subjective feelings of tension and apprehension, followed by autonomic nervous system responses at a given moment. Trait anxiety, assessed by the other scale, refers to a relatively stable tendency to perceive situations at threatening and react anxiously to them. The scores are divided into low, moderate, high and very high and are determined by the sum of 20 symptoms from a 5-point Likert-type scale.The range of scores is 20-80, the higher the score indicating greater anxiety for both the Trait and State Anxiety.
Time Frame: 90 days
Population: It was analysed only the number of participants that ended the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auriculotherapy Group | Control Group | Placebo Group
Number analyzed (Participants) | 24 | 25 | 22
units on a scale
  Trait Anxiety | 52.58 (9.29) | 49.48 (7.57) | 51.18 (10.32)
  State Anxiety | 54.04 (10.74) | 50.16 (10.79) | 51.59 (11.70)
Statistical Analysis 1: Comparison: Auriculotherapy Group vs Control Group vs Placebo Group; It was carried out the analysis of variance (ANOVA)of the medium difference among the groups in the 3rd (12 sessions) Hypothesis: there is at least one difference among the groups (State Anxiety); Test type: Superiority or Other; p = 0.012, ANOVA — After ANOVA it was performed Post Hoc Test and the statistical significance was p<0.05
Statistical Analysis 2: Comparison: Auriculotherapy Group vs Control Group vs Placebo Group; It was carried out the analysis of variance (ANOVA) of the medium difference among the groups at the follow-up (after 15 days). Hypothesis: there is at least one difference among the groups (State Anxiety); Test type: Superiority or Other; p = 0.005, ANOVA — After ANOVA, the Post Hoc Test was done and the statistical significance was p<0.05

ADVERSE EVENTS:
Time Frame: 3 months
Description: Tenderness and pain at the auricular point after the treatment
Arm/Group | Auriculotherapy Group | Control Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 1/24 | 0/25 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auriculotherapy Group (N=24) | Control Group (N=25) | Placebo Group (N=22)
Pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Pain and sensibility at the point after the treatment

LIMITATIONS AND CAVEATS:
The limitation of the trial was the reduced number of the sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The copyright of the search results are the exclusive property of the Journal of School Nursing, University of Saint Paul, barring any reproduction, in whole or in part in any form or means of printed or electronic, without the prior and necessary authorization is requested.